CLINICAL TRIAL: NCT02344329
Title: A Comparison of Total Contact Casting (TCC-EZ) Using Human Amnion Allograft (AmnioExcel) Versus Total Contact Casting (TCC-EZ) and Standard Wound Care in Treating Diabetic Foot Ulcers (TAD)
Brief Title: A Comparison of TCC-EZ Using Human Amnion Allograft vs TCC-EZ and Standard Wound Care in Treating Diabetic Foot Ulcers.
Acronym: TAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of North Dakota (Other)
Responsible Party: Principal Investigator, Patricia Thompson, Clinical Associate Professor, University of North Dakota
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TCC-104
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Diabetic Foot Ulcers; Diabetes
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus | interventions — Bandages

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): TCC-EZ and Standard Wound Care (Topical wound dressing) Two dressing and cast changes in week one followed by weekly applications until 12 weeks or closure which ever occurs first. Usual wound care would involve assessment, debridement, moist wound environment, and off-loading.
  Interventions: Device: Topical wound dressing; Other: usual wound care
- Intervention (Experimental): TCC-EZ and Human Amnion Allograft One dressing and two cast changes in week one followed by dressing change every two to three weeks and weekly cast changes until 12 weeks or closure which ever occurs first. Usual wound care would involve assessment, debridement, moist wound environment, and off-loading.
  Interventions: Biological: Human Amnion Allograft; Other: usual wound care

INTERVENTIONS:
Device: Topical wound dressing — Topical Wound Dressing
  Arms: Control
Biological: Human Amnion Allograft — Change dressing every two to three weeks and TCC-EZ is changed weekly for 12 or until healed.
  Other Names: AmnioExCel
  Arms: Intervention
Other: usual wound care — assessment, wound cleansing, debridement, moist wound environment, and off-loading

SUMMARY:
A Comparison of AmnioExcel® and Total Contact Casting (TCC-EZ) Versus Standard Wound Care and TCC-EZ in Treating Diabetic Foot Ulcers Best practice is to treat DFUs with standardized care and, if unsuccessful, use advanced modalities. This prospective clinical trial will compare healing rates between two treatment modalities in patients with DFUs in an ambulatory wound care clinic. The treatments are Total Contact Cast (TCC-EZ) with AmnioExcel® and TCC-EZ with standard treatment.

Adult participants 18 years or older with a diabetic foot ulcer located on the plantar surface and >1 cm in diameter will be asked by the Altru Wound Care Clinic MD or Family Nurse Practitioner visit to participate in the study if they have not demonstrated a 50% in reduction in wound area after two weeks of standard treatment. For those potential subjects who do not have 3rd party reimbursement the cost of the product and application will be covered by the respective company. They must be cognitively intact as evaluated by wound clinic primary care providers. Participants must agree to use the study treatments as directed, and to keep clinic visits during the 12-week trial or until the ulcer closes, whichever comes first.

DETAILED DESCRIPTION:
A TCC offloads pressure and is the gold standard for DFU treatment, as documented in several studies. The TCC results in an average healing rate of 80-90% within 6 weeks, yet only about 6% of DFU patients receive the TCC. The TCC requires special provider training for application. Given the high efficacy and low complication risk for the TCC, clinicians need to use the TCC to treat DFUs. Literature supports use of the TCC combined with other wound bed treatment modalities. AmnioExCel® is a dehydrated, extracellular human amnion derived tissue allograft that provides a structural tissue matrix that promotes angiogenesis, collagen matrix formation and re-epithelization (Werber et al., 2013). This study will look at whether or not combining AmnioExCel® and a TCC-EZ results in a better healing rate than TCC-EZ and standard wound care.

Purpose/Research Questions:

The purpose of this prospective clinical trial is to compare healing rates between two treatment modalities in patients with DFUs in an ambulatory wound care clinic. The treatments are Total Contact Casting (TCC-EZ) with AmnioExCel® and TCC-EZ with standard treatment.

Research Questions:

1. What is the difference in reduction in wound bed area for diabetic foot ulcers (DFUs) treated with Total Contact Casting TCC-EZ and AmnioExCel® compared to those treated with TCC-EZ and standard wound treatment?
2. What is the difference in time to closure for DFUs treated with TCC-EZ and AmnioExCel® compared to those treated with TCC-EZ and standard wound treatment?
3. What is the difference in cost of treatment for a diabetic foot ulcer treated with TCC-EZ and AmnioExCel® as compared to TCC-EZ with standard wound treatment?
4. What is the relationship between the hemoglobin A1c test(HbA1c) or glycated hemoglobin test and reduction in wound bed area for DFUs treated with TCC-EZ and AmnioExCel® compared to those treated with TCC-EZ and standard wound treatment?
5. What is the relationship between HbA1c and time to closure for DFUs with TCC-EZ and AmnioExCel® compared to those treated with TCC-EZ and standard wound treatment?
6. What is the subjects' reported satisfaction using TCC-EZ?
7. What is the reoccurrence of DFUs in a 90 day post treatment follow up?
8. What are the characteristics of adverse side effects using TCC-EZ and AmnioExCel®?

Methods:

All patients in this study will receive 2 weeks of usual wound care consisting of wound cleansing, removal of pressure (offloading), sharp debridement as needed, and maintenance of a moist wound environment. If they have demonstrated less than a 50% improvement in reduction in wound area of their DFU over 2 weeks, subjects will be approached for participation in this study. If they agree to participate, they will be randomly assigned to one of the two treatment groups. Treatment for Group A will consist of TCC-EZ® and AmnioExCel® and treatment for Group B will consist of standard wound care and TCC-EZ® and standard wound care. If the subject has more than one ulcer the largest ulcer will be used for inclusion in the study. At the beginning and end of the study blood samples for HbA1c will be taken and if the HbA1c is greater than 15%, subjects will be excluded or if random blood sugar is greater than 450 mg/dl (Marston et al., 2003). Study participation will be for 12 weeks or less if the wound closes before 12 weeks. DFUs not closed at the end of the 12 weeks of the study will continue to be treated until closed based on the decision of the Altru Wound Care Clinic providers. Complete wound closure will be defined as 100% re-epithelization without drainage or infection. Subjects clinic charts/records will be reviewed by the researchers to collect the following data: group assigned to, gender, age, diabetes diagnosis, co-morbidities, time ulcer has been present, if conventional treatment occurred for two weeks, date of 1st wound clinic visit, last HbA1c, date ulcer 1st noticed by patient, depth, and size of ulcer, ankle-brachial index, and ulcer characteristics at each visit will also be documented. At the conclusion of the study, subjects will complete a 12 question satisfaction questionnaire and six demographic questions on the TCC-EZ which will be administered by the clinic nurse or provider. Subjects may elect to withdraw from the study at any time without repercussion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be included if they are 18 years of age or older
* have a diagnosis of diabetes type 1 or 2
* random blood sugar of 450 or < and HbA1c of 15% or < drawn quarterly prior to study
* the ulcer has been present for a minimum of 2 weeks under the current investigators care
* the foot ulcer is on the plantar surface of the forefoot or heel and > 0.5cm2 in size at day 0
* patient's ulcer extends through the dermis into subcutaneous tissue but without exposure of bone or joint capsule classified as a grade 2 or 3 DFU using the University of Texas diabetic wound classification system
* ulcer is free of necrotic debris and appears to be made up of healthy vascularized tissue
* and subject's foot has evidence of adequate perfusion with an ankle-brachial index of > 0.7 and < 1.2.-

Exclusion Criteria:

* Subjects younger that 18 years of age
* no current diagnosis of diabetes type 1 or 2
* has uncontrolled hyperglycemia random blood sugar of > 450 mg/dl
* HbA1c > 15%
* gangrene present on any part of the affected foot
* ulcer's total surface area is > 20cm2
* ulcer has decreased or increased in size by 50% or more during the screening period
* presence of non-study ulcer located within 7.0 cm of the study ulcer at the beginning of the study day 0
* and evidence of infection determined by the provider.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-08; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Time to closure of a Diabetic Foot Ulcer using Human Amnion Allograft and Total Contact Casting vs Standard Wound Care and Total Contact Casting. | 12 weeks
  Number of days to closure of the DFUs.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A Thompson, MS,RN, Principal Investigator — University of North Dakota
Locations (1):
- Altru Health System, Grand Forks, North Dakota, United States

IPD SHARING:
Plan to Share IPD: Undecided